CLINICAL TRIAL: NCT01871662
Title: A Randomized, Single Center, Comparative Study to Evaluate the Efficacy and Safety of Silibinin (Legalon® SIL) in Combination With Ribavirin or With Peginterferon and Ribavirin, Versus Peginterferon and Ribavirin Based Standard of Care (SoC) in Treatment of naïve Genotype 4 Patients With Chronic Hepatitis C
Brief Title: Randomized Study for the Assessment of Silibinin (Legalon® SIL) in the Treatment of naïve Genotype 4 Patients With Chronic Hepatitis C
Acronym: HEPASIL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rottapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEG-SIL-2-02
Record Dates: First submitted 2013-05-30; First posted 2013-06-07 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C, Chronic
Keywords: HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Silybin; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group C: RIB + Peg-IFN (Active Comparator): Ribavirin(800-1400 mg/day,divided BID PO) + Peg-IFN alfa2b (1.5 μg/kg/week SC)for 25 weeks if RVR has been achieved or 49 weeks if EVR has been achieved
  Interventions: Drug: Pegylated interferon alfa2b; Drug: Ribavirin
- Group B:Legalon® SIL + RIB + Peg-IFN (Experimental): Silibinin (20 mg/Kg/day) for 6 days, followed by Silibinin + ribavirin (800-1400 mg/day, divided BID PO) + Peg-IFN alfa2b (1.5 μg/kg/week SC) for 15 days, followed by ribavirin (800-1400 mg/day, divided BID PO) + Peg-IFN alfa2b (1.5 μg/kg/week SC) + 2 days of Silibinin per week for 9 weeks, followed by ribavirin (800-1400 mg/day, divided BID PO) + Peg-IFN alfa2b (1.5 μg/kg/week SC) for 13 weeks if RVR has been achieved (for a total of 25 weeks of treatment) or 37 weeks if EVR has been achieved (for a total of 49 weeks of treatment)
  Interventions: Drug: Legalon® SIL (Silibinin); Drug: Pegylated interferon alfa2b; Drug: Ribavirin
- Group A: Legalon® SIL + RIB (Experimental): Silibinin (20 mg/Kg/day) for 6 days, followed by Silibinin + ribavirin (800-1400 mg/day, divided BID PO) for 15 days, followed by ribavirin (800-1400 mg/day, divided BID PO) + 2 days of Silibinin per week for 9 weeks, followed by ribavirin (800-1400 mg/day, divided BID PO) for 13 weeks if RVR has been achieved (for a total of 25 weeks of treatment) or 37 weeks if EVR has been achieved (for a total of 49 weeks of treatment)
  Interventions: Drug: Legalon® SIL (Silibinin); Drug: Ribavirin

INTERVENTIONS:
Drug: Legalon® SIL (Silibinin) — Silibinin 20 mg/Kg/day
  Arms: Group A: Legalon® SIL + RIB; Group B:Legalon® SIL + RIB + Peg-IFN
Drug: Pegylated interferon alfa2b — 1.5 µg/kg once-weekly
  Other Names: PEG-INTRON®
  Arms: Group B:Legalon® SIL + RIB + Peg-IFN; Group C: RIB + Peg-IFN
Drug: Ribavirin — At weight-based dose 800-1400 mg/day (BID, OS)
  Other Names: REBETOL®

SUMMARY:
The purpose of this study is to explore whether silibinin plus ribavirin with/without peg-interferon can be more effective than the peg-interferon plus ribavirin based standard of care (SoC) in the treatment of patients infected with hepatitis C virus genotype 4.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be willing to give written informed consent
* Male and female patients; age between 21 and 45 years inclusive
* Chronic hepatitis C infection with genotype 4 confirmed by genotypic testing at screening or within 6 months of screening period
* Patients eligible to be treated with RBV and Peg-IFN as per the instructions present in their prescribing information documents
* No history of prior interferon therapy (treatment naïve)
* Detectable HCV-RNA levels
* Normal BUN and creatinine
* Ability to communicate, participate, and comply with the requirements of the entire study

Exclusion Criteria:

* Liver transplant patients
* Co-Infection with HIV and/or HBV
* ALT >10-fold the upper limit of normal i.e. > 400 U/L
* Evidence of hepatocellular carcinoma (HCC)
* Fibroscan® at screening with a score ≥ 14.5 kPa
* Evidence of liver disease due to causes other than chronic HCV infection
* Evidence of poorly controlled diabetes (defined as HbA1c > 8%)
* History of alcohol or drug abuse within the last 12 months
* History or clinical evidence of liver decompensation, e.g. presence of ascites or encephalopathy, or bleeding from esophageal varices
* Serum albumin levels < 3.2 g/dL
* INR > 1.3 N
* Total Bilirubin levels > 2.0 mg/dL unless explained by Gilbert's disease
* Platelet Count < 100,000 µL
* Absolute Neutrophil counts < 1500 µL (mm3)
* Active or suspected non-hepatic malignancy or history of malignancy within the last 5 years
* Body Mass Index < 16 or > 35 kg/m2
* Females of childbearing potential:

  * Pregnancy (i.e. positive urine pregnancy test at screening) or lactation
  * Failure to agree to practice adequate contraception methods (e.g. oral contraceptives, intra-uterine device (IUD), transdermal contraceptive patch)
* Male patients not vasectomized, who do not agree to abstain from intercourse or who do not use a condom

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Undetectable HCV-RNA at 24 Weeks After the end of the Study Treatment | 24 weeks after the end of treatment (e.g. at week 49 or 73)
  The primary efficacy endpoint is the proportion of patients with Sustained Virological Response (SVR), i.e. undetectable HCV-RNA level lasting for 24 weeks after the completion of the study treatment course.

SECONDARY OUTCOMES:
Undetectable HCV-RNA | 4 weeks after the beginning of the study treatment
  Proportion of patients with Rapid Viral Response (RVR), i.e. undetectable HCV-RNA levels 4 weeks after the beginning of the study treatment course.
HCV-RNA decrease ≥ 2 log10 IU/mL | 12 weeks after the beginning of the study treatment
  Number and percentage of patients with Early Viral Response (EVR), i.e. HCV-RNA decrease ≥ 2 log10 IU/mL 12 weeks after the beginning of the study treatment course
Undetectable HCV-RNA | At the end of study treatment (e.g. at week 25 or 49)
  Proportion of patients with End Of Treatment (EOT) Response, i.e. undetectable HCV-RNA levels at the end of the study treatment (e.g. at the end of treatment at week 25 or 49)
Normalization of Serum Alanine Aminotransferase | 4 weeks after the beginning of study treatment, at EOT and at 24 weeks after the completion of the study treatment
  Proportion of patients with a normalization of Serum Alanine Aminotransferase (ALT <40 U/L) values 4 weeks after the beginning of study treatment, at EOT and at 24 weeks after the completion of the study treatment course;
Number of Participants with adverse events (AEs) | Up to 24 weeks after the end of treatment (e.g. up to week 49 or 73)

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Esmat, MD, Principal Investigator — Al-Manial University Hospital, Kasr El-Aini Faculty Medicine, Cairo University, Egypt; Samer El-Kamary, MD, Study Chair — University of Maryland School of Medicine,Baltimore, USA
Locations (1):
- Al-Manial University Hospital, Kasr El-Aini Faculty Medicine, Cairo University, Cairo, Egypt